CLINICAL TRIAL: NCT03273634
Title: The Effect of Proton Pump Inhibition on Palpitations With no Apparent Cause. A Double Blinded Randomized Placebo Controlled Trial
Brief Title: The Effect of Proton Pump Inhibition on Palpitations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jordan Collaborating Cardiology Group (Other)
Collaborators: University of Jordan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2017-08-21; First posted 2017-09-06 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Arrhythmia
Keywords: Palpitations
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Similarly looking tablets and placebo with care providers not knowing which is which. Packets are marked "heads and tails" for randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): The treatment will consist of lanzoprazole 30 mg once daily at night time
  Interventions: Drug: Lansoprazole Pill
- Placebo (Placebo Comparator): A Placebo pill to be given with similar looking to experimental drug but contains inactive ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lansoprazole Pill — once daily at night time
  Other Names: Lanzotec
  Arms: Active treatment
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Feeling of palpitations with no clear arrhythmia is frequently encountered in clinical practice. The majority of these patients have documented sinus rhythm even while having symptoms. Gastrointestinal association with such symptoms was first described by Ludwig von Roemheld (1871-1938).The investigators thought to investigate the effect of proton pump inhibition in patients with feeling of palpitations but no clear cause.

DETAILED DESCRIPTION:
One hundred and fifty patients with palpitations and no clear cause for their symptoms will be randomized to receive either proton pump inhibitor (PPI) (lanzoprazole 30 mg) or placebo for one month. At base line they will be investigated to rule out arrhythmia by documenting normal heart rate (less than 110 beat per minute) or ECG showing normal sinus rhythm or mild sinus tachycardia (Less than 110 per minute) during symptoms. Obvious causes such as anxiety due to a stressful event or organic causes such anemia or thyroid disorders should be also ruled out.

Patient who agree to participate in the study will be asked to sign an informed consent. A baseline questionnaire with symptoms will be filled. They will then be randomized for treatment with either PPI or placebo once at night time. After 10 days of treatment they will be contacted and questioned regarding their symptoms. The two groups will be compared to see if there is any improvement of symptoms with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with palpitations and no clear cause who are above the age of 16 years and who consent to the study will be included
2. Clear causes that should be excluded are true arrhythmia such SVT or VT or frequent premature atrial or ventricular contractions or any organic cause such as thyroid disorder, anemia (hg less than 11 g/dl) and obvious anxiety disorder
3. Arrhythmia can be excluded by an ECG showing sinus rhythm or sinus tachycardia during episodes or measurement of heart rate by a reliable method during symptoms showing regular heart rate less than 120 beats per minute.

Exclusion Criteria:

1. Refusal to sign consent form
2. Already taking PPI or H2 blocker
3. Frequency of symptoms less than 2 times per week

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Improvement in symptoms | 10 days after starting treatment
  Assessment of improvement in palpitations using a questionnaire. The improvement will be graded either non, mild, moderate, or great. The result will either negative (no or mild improvement), or positive (moderate or great improvement)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ubaidat, MD, Study Chair — Jordan University Hospital
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No